CLINICAL TRIAL: NCT04714580
Title: Traduzione e Validazione Italiana Del Protocollo di Esercizi Animal Fun
Brief Title: The Animal Fun Program to Support the Motor Development of the Italian Pre-schoolers: a Case-Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Francesca Policastro, Lecturer, PhD, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 86-7/3/2018 pg 6
Record Dates: First submitted 2021-01-07; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal Fun Group (Experimental): Baseline assessment with MABC-2; Animal Fun activity with a certified trainer (physiotherapist) for one month, three times a week, for 30 minutes; one-month follow-up assessment with MABC-2.
  Interventions: Other: Animal Fun Program
- Control Group (No Intervention): Baseline assessment with MABC-2; normal curricular activity at school with the teachers; one-month follow-up assessment with MABC-2.

INTERVENTIONS:
Other: Animal Fun Program — This program permits the operators to propose different activities, by following the needing of the children. As the name of this program suggests, all the activities involve an animal description, and ask the children to move like this animal, in a proper, correct and supervised way.
  Arms: Animal Fun Group

SUMMARY:
The present literature supports the importance of the motor activity since the early stages of the human development. The children with poor motor skills are at greater risk for psychosocial, internalizing, and metabolic diseases. In Italy data about obesity and inactivity are increasing, anyway there is lack of motor program for pre-schoolers. The movement program Animal Fun seems to be a valid tool to support these children. The aim of this study is to verify the feasibility of using Animal Fun with Italian pre-schoolers.

119 preschool children (3-6 years old) from 3 Italian kindergartens were included in this study. The schools were randomly allocated to intervention and control group. Movement Assessment Battery for Children - 2 (MABC-2) was administered to all the children at the baseline and at one-month follow-up. During this month, the schools assigned to the control group followed the normal curriculum; the schools assigned to the Animal Fun group, followed the Animal Fun activity (thirty minutes, thrice a week).

The investigators expect that the Animal Fun program demonstrates valid and feasible even in the Italian context, where there is lack of movement program supporting the development of the pre-school children.

DETAILED DESCRIPTION:
Rationale and Background:

Motor skills and physical activity are strongly related to the cognitive, physical, social and psychological development of children. They are also crucial in the prevention of cardiovascular or metabolic diseases, such as obesity or diabetes. There is growing evidence indicating that children with poor motor coordination may be at significant risk for psychosocial and internalizing problems. Other research has found significant levels of anxiety and depression even in 4-5-years-old-children.

Due to fear of failure, or of peer bullying, children with motor difficulties often limit their opportunity to practice motor activities, thus creating a vicious cycle. In this continuous negative loop, the child has low motor competency, develops low fitness training and tends towards hypo-activity. In contrast, if children are confident with their motor skills, they are more likely to participate in activities such as sports or dancing. Literature also relates the motor ability of preschool children to their scholastic adaptation and to the social adjustment in the first year of school.

Preschool is an essential period in a child's life because Fundamental Movement Skills are developing at this stage, for both gross and fine motor tasks.

Some investigators have demonstrated that most pre-schoolers don't practice the recommended amount of daily physical activity. Unfortunately, there is a lack of movement programs to engage pre-school children in motor activities. In 2010, the Curtin University developed the "Animal Fun" program. This program was designed to provide developmentally appropriate activities that would be fun and engaging for all children aged 3-6 years whilst targeting specific areas of development. They created a protocol, which will benefit all children in the group - those with and without motor difficulties. By referring to all the members of a class, Animal Fun avoids the stigma associated with "special programs". This is an ecological program for use in schools during the ordinary activities. Animal Fun is an imaginative program of movement, in which the children imitate animals' movements. It is flexible and doesn't provide a rigid structure to follow, but it adapts to children's interests and abilities. Evidence demonstrates, that Animal Fun supports the development of overall motor ability, particularly throwing and balance skills, and significantly improves social skills in young children.

In Italy there is a lack of motor programs for pre-schooler children. Furthermore, children with poor motor skills are not recognized, therefore no specific support is provided. The need to identify an inclusive and flexible motor program has led us to Animal Fun. Considering the socio-cultural differences between Western Australia and Italy, the purpose of this study is to verify the feasibility of the Animal Fun program for Italian pre-schoolers. Study goals and objectives:

In Italy there is lack of motor program for pre-schoolers, like Animal Fun. The first aim of this study is understanding the feasibility of this activity in the Italian kindergartens. Second, this study would understand the validity of the results of one month of Animal Fun practice. Using the gold standard assessment for motor skills in children, Movement Assessment Battery for Children - 2 (MABC-2), the main objective is to verify the motor improvements in children who practiced Animal Fun, compared to a control group. This assessment provides score about the manual dexterity, the balance and the aiming and catching skills. A sum of these scores provides a total score about the motor skills, in general. Through this test, understanding the motor competences of the pre-schoolers is affordable.

Study design:

This study is a longitudinal randomized controlled trial, and it is participants' blinded.

It has been approved from the Ethics Committee of the University of Trieste. All methods were performed in accordance with the relevant guidelines and regulations, especially the Helsinki Declaration.

As first, kindergartens' directors gave the consent to participate in the study.

3 Kindergartens of the province of Trieste have been recruited and randomly allocated to Animal Fun intervention (1), and control group (2). From the three schools, we recruited 119 pre-schoolers. The parents previously read and signed the written informed consent, to let the child participating.

Inclusion criteria: written informed consent, attending one of the three involved kindergartens, 3-6 years old.

Exclusion criteria: not-typically developing children and children with specific sickness.

The duration of the study is two months.

Methodology:

As first, all the parents informed the investigators about the specific age of the child, the hand preference, and the presence of such a deficit or disease. These data were necessary to set up the assessment for each child. In fact, some administration-differences exist, especially between ages.

Intervention group: baseline assessment with MABC-2; Animal Fun activity with a certified trainer (physiotherapist) for one month, three times a week, for 30 minutes; one-month follow-up assessment with MABC-2.

Control group: baseline assessment with MABC-2; normal curricular activity at school with the teachers; one-month follow-up assessment with MABC-2

Animal Fun activity was carried out following all the instructions given by the authors in the published book. This program permits the operators to propose different activities, by following the needing of the children. The proposed activities are entirely described in the nine modules of this tool.

Before the assessment, the investigators decided to use 30 motor activities (on 97 available) with the intervention group. As the name of this program suggests, all the activities involve an animal, and ask the children to move like this animal, in a proper, correct and supervised way.

After the assessment, considering the mean-scores of the children and their percentiles, the investigators decided to focus especially on the activities for improving the balance, and the aiming and catching skills. In fact, the children scored lower in these activities then in the manual dexterity test. For this, most of the activities of the first modules of Animal Fun have been proposed, which focus on the balance on two/one foot, on the locomotion, on the balance during a throw, on the aim. The animals involved were, for instance, the flamingo, the elephant, the dog, the monkey, and more.

To the teachers of the control group, the investigators gave no additional information about what to do during the curricular activities, in order no to create a bias. Even the teachers of this group were blinded about the study.

Safety considerations:

In this study, the safety of the participants was guarantee. All the activities of the intervention group were coordinated and managed by a certified trainer, who could control the safety of the children during Animal Fun. Every possibile accident during the motor activity was considered as normal accident during the kindergarten time, and consequently managed by the teachers. The parents were previously informed about this issue, in the written informed consent.

Follow-up:

After the second assessment with the MABC- 2 at one-month follow-up, the participants are followed no more from the researchers of the present study.

Data management and statistical analysis:

Analysis was conducted in R (R Core Team, 2017) and graphs were produced using the package Rcmdr and its plug-ins.

Normality of the variables was assessed through Shapiro-Wilk test. Intervention and control groups were compared at the baseline through Fisher test for the qualitative variables, and through the t-test for the quantitative ones. The time Δt was created to define the difference between the final and the basal scores. The two groups were compared considering Δt through the Mann-Whitney test. Kaplan-Meier estimate of the median, and 95% confidence interval were reported for each variable at Δt.

Expected outcomes of the study:

The outcomes of this study could be very significant considering the possibility of introducing Animal Fun in the Italian kindergartens, as curricular motor activity. The impact of this program of movement on the quality of the life of the pre-schoolers can be huge. Furthermore, giving the possibility to these children to move, and learn, can also give a benefit considering the prevention of metabolic, cardio-vascular, postural and psycho-social diseases.

This project didn't received any fund, budget or sponsor's support.

ELIGIBILITY:
Inclusion Criteria:

* parents written informed consent
* attending one of the three involved kindergartens
* 3-6 years old.

Exclusion Criteria:

* not-typically developing children
* children with specific sickness

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change form Baseline Movement Assessment Battery for Children-2 at 1 month follow-up | One month
  This test is suitable for children and adolescents aged 3 to 17 years, and assesses the motor skills of children in the following domains: Aiming and Catching (AC), Balance (Bal), and Manual Dexterity (MD). Cluster and total standard scores for children are provided, with higher scores demonstrating better performance. A total test score (Tot MABC-2) at or below the 5th percentile indicates significant movement difficulty, while a score between the 5th and 15th percentile indicates that a child is "at risk".
  In these tests, the items and the scores were compared to the normative data of the uploaded version of the Italian MABC-2.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Policastro, PhD, Principal Investigator — Univerisity of Trieste
Locations (1):
- University of Trieste, Physiotherapy Degree, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No
Each family will receive a summary of the results of assessment, in order to make them aware of the motor skills.
  Other researcher will be able to consult the complete results of the study and the study protocol.

REFERENCES:
- [Background] Piek JP, Straker LM, Jensen L, Dender A, Barrett NC, McLaren S, Roberts C, Reid C, Rooney R, Packer T, Bradbury G, Elsley S. Rationale, design and methods for a randomised and controlled trial to evaluate "Animal Fun"--a program designed to enhance physical and mental health in young children. BMC Pediatr. 2010 Nov 4;10:78. doi: 10.1186/1471-2431-10-78. PMID 21050483
- [Background] Piek JP, Kane R, Rigoli D, McLaren S, Roberts CM, Rooney R, Jensen L, Dender A, Packer T, Straker L. Does the Animal Fun program improve social-emotional and behavioural outcomes in children aged 4-6 years? Hum Mov Sci. 2015 Oct;43:155-63. doi: 10.1016/j.humov.2015.08.004. Epub 2015 Aug 27. PMID 26298689
- [Background] Piek JP, McLaren S, Kane R, Jensen L, Dender A, Roberts C, Rooney R, Packer T, Straker L. Does the Animal Fun program improve motor performance in children aged 4-6 years? Hum Mov Sci. 2013 Oct;32(5):1086-96. doi: 10.1016/j.humov.2012.08.004. Epub 2012 Nov 24. PMID 23186610
- [Background] De Oliveira JA, Rigoli D, Kane R, McLaren S, Goulardins JB, Straker LM, Dender A, Rooney R, Piek JP. Does 'Animal Fun' improve aiming and catching, and balance skills in young children? Res Dev Disabil. 2019 Jan;84:122-130. doi: 10.1016/j.ridd.2018.07.004. Epub 2018 Aug 4. PMID 30087016
- See also: Website of Animal Fun Program — https://animalfun.com.au